CLINICAL TRIAL: NCT06518499
Title: Outcomes of Karydakis, Primary Closure, and Pit Picking Methods in the Treatment of Pilonidal Sinus: A Prospective Study in Women
Status: Recruiting | Type: Observational
Sponsor: Sehit Prof. Dr. Ilhan Varank Sancaktepe Training and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Ivstrh 172
Record Dates: First submitted 2024-07-12; First posted 2024-07-24 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-07

CONDITIONS: Pilonidal Sinus
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Bascom's Pit-Pick procedure: The Bascom pit-pick procedure is performed under local anesthesia with the patient in a prone position, taking approximately 15-20 minutes. Pre-operative preparation includes shaving and cleaning the surgical area. Local anesthesia (lidocaine with adrenaline) is typically used, with general anesthesia as an alternative if needed. The surgical technique involves excising midline pits with a scalpel, removing infected granulation tissue and hairs through curettage or a lateral incision. Midline wounds and nearby secondary pits are sutured with polypropylene, while the lateral incision is left open and covered with a hydrofibre bandage to heal by secondary intention.
  Interventions: Procedure: Pilonidal sinus surgery
- Primary Closure: The primary closure technique for pilonidal sinus involves placing the patient in a prone position under spinal or general anesthesia, shaving and cleaning the surgical area, and making an elliptical incision to remove the affected tissue. A skin flap is then mobilized from the surrounding area to cover the excision site, and the wound is closed with sutures.
  Interventions: Procedure: Pilonidal sinus surgery
- Karydakis: The Karydakis primary closure procedure involves placing the patient in a prone position under spinal or general anesthesia. The surgical area around the natal cleft is shaved and cleaned thoroughly. A symmetric elliptical excision is performed 2 cm lateral to the midline, removing all affected pilonidal sinus tissue and some surrounding normal tissue. A skin flap, 2 cm wide and 1 cm thick, is mobilized from the contralateral side to cover the resultant defect. The flap is secured using a continuous suture technique, with the skin closed using polypropylene mattress sutures. A low-suction drain is used to standardize the procedure, removed when drainage decreases to less than 20 ml/day.
  Interventions: Procedure: Pilonidal sinus surgery

INTERVENTIONS:
Procedure: Pilonidal sinus surgery — Bascom's Pit-Pick procedure, Primary Closure, Karydakis procedure

SUMMARY:
Although there are many methods for the surgical treatment of pilonidal sinus disease, the number of studies specific to women is limited in the literature. In addition to post-treatment recurrence and complication rates in women, aesthetic results are also of great importance. This study will compare the Karydakis procedure, a flap method, and the Bascom's pit-pick procedure, a minimally invasive procedure, in terms of recurrence, complications and aesthetics, especially in female patients with three or fewer pits.

DETAILED DESCRIPTION:
This study is a single-center, prospective observational trial aimed at comparing the effectiveness of the Karydakis flap and Bascom's pit-pick methods in treating pilonidal sinus disease in women. Female patients aged 18 and over, with three or fewer pits, will be included, and each patient will be followed for 12 months. The Bascom pit-pick method will be performed under local anesthesia, while the Karydakis method will be performed under spinal or general anesthesia. Postoperative recovery time, complications, recurrence rates, and patient satisfaction will be evaluated. Ethics committee approval has been obtained (Approval No: TE 172, Date: June 12, 2024).

ELIGIBILITY:
Inclusion Criteria:

* Female patients 18 years old and older
* Diagnosed with pilonidal sinus disease, having 3 or fewer pits.
* No previous surgical treatment for pilonidal sinus.

Exclusion Criteria:

* Under 18 years of age
* Pregnancy
* Presented with acute abscesses
* Patients with recurrent disease, Stage-R.
* >3 pit
* Collagen tissue disease
* Exceed to navicular area
* Lateral extension in both directions
* Accidentally discovered (asymptomatic) sinus or with follow-up <12 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Female patients aged 18 and older with pilonidal sinus disease and three or fewer pits, with no previous surgical treatment.
Sampling Method: Probability Sample
Enrollment: 145 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-20 (Estimated)

PRIMARY OUTCOMES:
Recurrence Rate | 12 months post-surgery
  This measure evaluates the rate of pilonidal sinus disease recurrence in female patients undergoing Karydakis flap or Bascom's pit-pick surgical procedures over a 12-month period. Recurrence is defined as the reappearance of disease symptoms after the wound has completely healed.

SECONDARY OUTCOMES:
Complication Rate | 30 days post-surgery
  This measure records the incidence of postoperative complications such as infections (superficial or deep), seromas, hematomas, wound dehiscence (partial or complete), and anesthesia-related complications within the first 30 days post-surgery.
Aesthetic Outcome (Visual Analog Score for pain) | Up to 1 year post-surgery
  Assessment of aesthetic outcomes using the Visual Analog Scale (VAS) for pain. The VAS is a scale from 0 to 10, where 0 represents no pain and 10 represents the worst possible pain. Higher scores indicate worse outcomes.
Healing Time | Up to 12 weeks post-surgery
  This measure records the time required for complete wound healing post-surgery, defined as the integrity along the incision line without any complications.
Functional Recovery | Up to 24 weeks post-surgery
  This measure assesses the time taken for patients to resume daily activities comfortably.

CONTACTS AND LOCATIONS:
Locations (1):
- Sancaktepe Sehit Prof. Dr. Ilhan Varank Training and Research Hospital, Istanbul, Other, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol